CLINICAL TRIAL: NCT05843500
Title: Chronic Thromboembolic Disease: A Prospective Registry
Brief Title: Chronic Thromboembolic Disease Registry
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 23-38534
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Chronic Thromboembolic Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic thromboembolic disease: Patients with chronic thromboembolic disease/pulmonary hypertension
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients who received medical, surgical or interventional treatment for chronic thromboembolic pulmonary hypertension will be followed and given quality of life questionnaires.

SUMMARY:
The goal of this patient registry is to learn about the natural history in patients with chronic thromboembolic disease (CTD) and/or chronic thromboembolic pulmonary hypertension (CTEPH). The main question[s] it aims to answer are:

* Long-term outcome after various types of treatment, including medication, balloon pulmonary angioplasty, and pulmonary endarterectomy
* Effect of treatment on patient's quality of life and exercise tolerance Participants will be followed longitudinally to assess their health outcomes and quality of life via chart review and health quality surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred with CTED and/or CTEPH defined as:

  1. Mean pulmonary arterial pressure (mPAP) > 20 mmHg at rest with pulmonary vascular resistance (PVR) > 2 Wood units (WU); or if mPAP ≤ 20 mmHg or PVR ≤ 2 WU at rest, have exercise limitations from chronic thromboembolic pulmonary disease (CTEPD) without pulmonary hypertension (PH)
  2. Radiologic finding of chronic thromboembolic disease, including abnormal ventilation perfusion scan, pulmonary angiogram, computer tomographic pulmonary angiogram, or magnetic resonance pulmonary angiogram
  3. Post-embolic exercise intolerance and evidence of chronic thromboembolic disease in the absence of resting pulmonary hypertension
* Treatment with anticoagulation for ≥ 3 months before diagnosis of CTEPH or CTEPD without PH
* Age ≥ 18 years

Exclusion Criteria:

* Main cause of PH other than World Health Organization (WHO) group 4 (CTEPH)
* Patient's refusal to participate in clinical research and/or receive intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed chronic thromboembolic disease (CTED) or chronic thromboembolic pulmonary hypertension (CTEPH)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Total number of patients who survive | Through study completion, an average of 5 years
  The total number of patients who are alive
Changes in exercise tolerance | Baseline to end of the study, an average of 5 years
  Measured by 6-min walk test, which will be done approximately every 3 months at follow up per standard of care
Changes in supplemental oxygen use severity | Baseline to end of the study, an average of 5 years
  Number of patients on supplemental oxygen, which will be recorded approximately every 3 months at follow up per standard of care. This will be compiled at the end of the study to provide overall change in measurement.
Changes in New York Heart Association (NYHA) functional class | Baseline to end of the study, an average of 5 years
  Grading of patients by NYHA functional class, which include functional capacity and objective assessment. This will be compiled at the end of the study to provide overall change in measurement.
European Quality of Life Five Dimension (EQ-5D) - Scale Score | Baseline to end of the study, an average of 5 years
  Assessment of quality of life will be measured using EQ-5D-5L. This instrument is a self-assessed, health-related, quality of life questionnaire that measures quality of life on a 5-component scale. The scores range from Level 1 to Level 5, with lower scores indicating a higher quality of life. This will be collected every 3 months and compiled at the end of the study to provide overall change in measurement.
Changes in patients' emPHasis-10 scores | Baseline to end of the study, an average of 5 years
  Assessed by the emPHasis-10 (pulmonary hypertension) instrument, which is an instrument specifically designed to assess the quality of life in patients with pulmonary hypertension. Each item will be scored from 0 to 5 where 0 was the best score. This will be collected every 3 months and compiled at the end of the study to assess overall change in measurement.
Number of patients undergoing lung transplantation | Baseline to end of the study, an average of 5 years
  Number of patients undergoing lung transplantation

SECONDARY OUTCOMES:
Changes in CTEPH-/CTED- specific medication | Baseline to end of the study, an average of 5 years
  The frequency and dose of medication specifically for management of CTEPH or CTED, which will be assessed approximately every 3 months as routine medical follow up. This will be compiled at the end of the study to assess overall change.
History of undergoing pulmonary endarterectomy | Through study completion, an average of 5 years
  Number of patients undergoing pulmonary endarterectomy
History of undergoing pulmonary balloon angioplasty | Through study completion, an average of 5 years
  Number of patients undergoing pulmonary balloon angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Miles Conrad, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No